CLINICAL TRIAL: NCT00138866
Title: Risedronate for Treatment of Sublesional Osteoporosis After Spinal Cord Injury
Brief Title: Risedronate for the Treatment of Osteoporosis for People With Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); St. Joseph's Health Care London (Other)
Responsible Party: Dr. BC Craven, Toronto Rehab Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRI REB #04-016; PSI #03-52
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2008-07

CONDITIONS: Osteoporosis
Keywords: Spinal cord injury
MeSH Terms: conditions — Osteoporosis; Spinal Cord Injuries | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Risedronate

SUMMARY:
The purpose of this study is to find out if risedronate works for the treatment of osteoporosis for people with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury of greater than 18 months
* Osteopenia or osteoporosis of the hip
* Must be able to swallow tablets and sit upright

Exclusion Criteria:

* Bilateral heterotopic ossification
* Bilateral lower extremity metal implants
* Pregnant or lactating females
* Paget's disease
* Osteomalacia
* Steroid induced bone loss
* Untreated parathyroid or thyroid disease
* Symptomatic hypocalcemia or hypophosphatemia
* Treatment in the last year with calcitonin, fluoride or anabolic steroids
* Current treatment with prednisone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2004-11; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density of the distal femur between baseline and 18-months | 18 months

SECONDARY OUTCOMES:
Change in bone mineral density of the hips and proximal tibia between baseline and 18-months | 18 months
The change in biochemical bone markers of bone turnover between baseline and 18-months | 18 months
The frequency and severity of adverse events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: B. Cathy Craven, MD, FRCPC, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehab, Lyndhurst Centre, Toronto, Ontario, Canada